CLINICAL TRIAL: NCT05804461
Title: Optimizing PrEP Uptake Among Latino MSM in Puerto Rico: A Comparative Effectiveness Study
Brief Title: Optimizing Pre-Exposure Prophylaxis (PrEP) Among Latino Men Who Have Sex With Men (MSM) in Puerto Rico
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2290030276
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face intervention (Experimental): A three-session face-to-face intervention using Motivational Interviewing with a facilitator; to increase Pre-Exposure Prophylaxis (PrEP) uptake. Pre-post-post evaluations after each session will be administered. Participation will last 150 days from the start to the last follow-up.
  Interventions: Behavioral: Motivational Interviewing
- Online intervention (Experimental): A three-session online intervention using Motivational Interviewing with a facilitator; to increase Pre-Exposure Prophylaxis (PrEP) uptake. Pre-post-post evaluations after each session will be administered. Participation will last 150 days from the start to the last follow-up.
  Interventions: Behavioral: Motivational Interviewing
- Control (No Intervention): No intervention. Pre-post evaluations will be administered.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Upon refinement from Formative Research (Aim 1), a three-session, individual-level intervention to increase Pre-Exposure Prophylaxis (PrEP) uptake among men who have sex with men (MSM) in Puerto Rico will be implemented. The facilitator will use Motivational Interviewing techniques to guide the sessions. The intervention's design and content will be the same for each study group; the only difference will be the modality of implementation; one group of participants will receive a face-to-face intervention, while another group will receive an online intervention.A total of 170 participants will be randomized in a 1:1 ratio into each of the two intervention modalities (n=85 face-to-face and n=85 online) while a control group will be recruited following a 3:1 ratio of intervention vs. control. In addition to baseline assessment, participants will be asked to complete a post test at the end of the third session (60 days) and a follow-up post-test at the 150-day mark, separately.
  Arms: Face-to-face intervention; Online intervention

SUMMARY:
To develop, assess and compare the effectiveness of a Motivational Interviewing Intervention for increasing Pre-Exposure Prophylaxis (PrEP) uptake among Latino Men Who Have Sex With Men (MSM) in Puerto Rico.

ELIGIBILITY:
Latino MSM group - Inclusion Criteria:

* Biological male
* Age 21 or older
* Self-reported HIV negative or unknown status
* Not using PrEP (participants who have discontinued PrEP use can participate in the study), Spanish fluency (ability to write and read in Spanish)
* Presenting at least one of the eligibility criteria for PrEP as established by the CDC (including men who have had an infection (STI) in the past 6 months, HIV positive sexual partner)
* Access to a portable technology device (e.g., phone, tablet, laptop) or desktop computer access to internet connection

Exclusion Criteria:

* HIV positive individual
* Evidence of being under the effects of alcohol or drugs
* Indication of unstable or serious psychiatric symptoms
* Evidence of major cognitive impairment
* Inability to speak and read in Spanish

Healthcare Providers group - Inclusion Criteria:

* Age 21 or older
* Providing PrEP related health services at time of enrollment (e.g., case management, clinical services)
* Spanish fluency (ability to write and read in Spanish)

Exclusion Criteria:

* Evidence of being under the effects of alcohol or drugs
* Indication of unstable or serious psychiatric symptoms
* Evidence of major cognitive impairment
* Inability to speak and read in Spanish

Ages: 21 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary | 150 days
  PrEP uptake

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided